CLINICAL TRIAL: NCT06130202
Title: Echocardiographic Findings as Markers of Subclinical Cardiac Dysfunction in Patients With Non-Alcoholic Fatty Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Mohamed Abdel-Naiem Mossad, Principale Investigator, Assiut University
Other Study IDs: Echocardiographic in NAFLD
Record Dates: First submitted 2023-10-20; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-10

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NAFLD
  Interventions: Device: Echocardiographic findings

INTERVENTIONS:
Device: Echocardiographic findings — Echocardiographic findings as Markers of Subclinical Cardiac dysfunction in Patients with Non-Alcoholic Fatty Liver Disease

SUMMARY:
The investigators aim to evaluate patients with NAFLD for early echocardiographic signs of myocardial dysfunction and if there is any correlation between the degree of steatosis or fibrosis and the degree of myocardial dysfunction. This might be an early predictor for anticipating cardiac dysfunction in such cases who are naturally at more increased risk of cardiovascular complications.

DETAILED DESCRIPTION:
Individuals with Non-Alcoholic Fatty Liver Disease (NAFLD) have abnormal myocardial energy metabolism and reduced coronary functional capacity, even in the absence of risk factors for cardiovascular disease (CVD) ,Nonalcoholic fatty liver disease (NAFLD) is now recognized as the most common cause of chronic liver disease worldwide , Its prevalence has increased to more than 30% of adults in developed countries and its incidence is still rising , The majority of patients with NAFLD have simple steatosis but in up to one third of patients, NAFLD progresses to its more severe form nonalcoholic steatohepatitis (NASH) , NASH is characterized by liver inflammation and injury thereby determining the risk to develop liver fibrosis and cancer , NAFLD is considered the hepatic manifestation of the metabolic syndrome. However, the liver is not only a passive target but affects the pathogenesis of the metabolic syndrome and its complications. Conversely, pathophysiological changes in other organs such as in the adipose tissue, the intestinal barrier or the immune system have been identified as triggers and promoters of NAFLD progression , Metabolic syndrome is a cluster of metabolic abnormalities that identifies people at risk of diabetes and cardiovascular disease, whereas non-alcoholic fatty liver disease (NAFLD) is defined as a disorder with excess fat in the liver due to non-alcoholic causes. Two key components of metabolic syndrome, glucose and triglycerides, are overproduced by the fatty liver. The liver is therefore a key determinant of metabolic abnormalities. The prevalence of both metabolic syndrome and NAFLD increases with obesity. Both disorders predict type 2 diabetes, cardiovascular disease, non-alcoholic steatohepatitis (NASH), and hepatocellular carcinoma , Because metabolic syndrome can be defined in many different ways, NAFLD might be a more direct predictor of these diseases , Several cohort studies have consistently documented that NAFLD (especially in its more advanced forms) is associated with a higher risk of all-cause mortality and that the leading causes of death among patients with NAFLD are cardiovascular diseases (CVDs), followed by extrahepatic malignancies and liver-related complications , A growing body of evidence also indicates that NAFLD is strongly associated with an increased risk of major CVD events and other cardiac complications (ie, cardiomyopathy, cardiac valvular calcification and cardiac arrhythmias), independently of traditional cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* all NAFLD patients who will be seen in the outpatient clinic in our hospital. Diagnosis of NAFLD will be based on clinical history and examination, imaging and fibroscan results

Exclusion Criteria:

1. Children less than 16 years
2. Adults more than 70 years
3. Known advanced cardiovascular disease as:

   * advanced heart failure with reduced ejection fraction (HFrEF)
   * history of recent acute myocardial event as acute coronary syndrome
   * symptomatic chronic myocardial ischemia
   * Known or recent diagnosis of rheumatic heart disease
   * Known or recent diagnosis of congenital heart disease
4. Advanced comorbidities: advanced cancer, chronic kidney disease, advanced liver disease (decompensated cirrhosis), and advanced pulmonary disease.

Ages: 17 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: -Study tools (in detail, e.g., lab methods, instruments, steps, chemicals,): all participants will be subjected to full history taking and examination with attention to inclusion and exclusion criteria and other comorbidities as follows:
  * Clinical evaluation: for:
    * history and possible etiology of NAFLD
    * confirming inclusion and exclusion criteria
    * Body weight and height, and body mass index (BMI)
  * Lab investigations:
    1. complete blood count
    2. liver function tests
    3. coagulation profile (PT - PC - INR)
    4. kidney function tests (urea, creatinine and e-GFR)
    5. HBA1C
    6. Complete lipid profile (total cholesterol, LDL, HDL and Triglycerides)
    7. Serum TSH
    8. electrolytes (Na, K, Calcium, MG, PO4)
  * Imaging:
    * Abdominal us
    * Fibroscan to assess liver stiffness (LSM) graded from F0 to F4 and degree of steatosis using the CAP score
    * 2-D conventional transthoracic echocardiography
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2023-11-20 (Estimated); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
evaluate patients with NAFLD for early ECHOCARDIOGRAFPHIC signs of MYOCARDIAL DYSFUNCTION . | through study completion, an average of 1 year
  Patient outcomes will be recorded and analyzed. Statistical analysis will be done using measures of correlation and regression using up-to-date statistical analysis tools.

SECONDARY OUTCOMES:
if there is any CORRELATION between the degree of STEATOSIS or FIBROSIS and the degree of MYOCARDIAL DYSFUNCTION . | through study completion, an average of 1 year
  Patient outcomes will be recorded and analyzed. Statistical analysis will be done using measures of correlation and regression using up-to-date statistical analysis tools

REFERENCES:
- [Background] Younossi ZM, Koenig AB, Abdelatif D, Fazel Y, Henry L, Wymer M. Global epidemiology of nonalcoholic fatty liver disease-Meta-analytic assessment of prevalence, incidence, and outcomes. Hepatology. 2016 Jul;64(1):73-84. doi: 10.1002/hep.28431. Epub 2016 Feb 22. PMID 26707365
- [Background] Saab S, Manne V, Nieto J, Schwimmer JB, Chalasani NP. Nonalcoholic Fatty Liver Disease in Latinos. Clin Gastroenterol Hepatol. 2016 Jan;14(1):5-12; quiz e9-10. doi: 10.1016/j.cgh.2015.05.001. Epub 2015 May 11. PMID 25976180
- [Background] Pan JJ, Fallon MB. Gender and racial differences in nonalcoholic fatty liver disease. World J Hepatol. 2014 May 27;6(5):274-83. doi: 10.4254/wjh.v6.i5.274. PMID 24868321
- [Background] Fleischman MW, Budoff M, Zeb I, Li D, Foster T. NAFLD prevalence differs among hispanic subgroups: the Multi-Ethnic Study of Atherosclerosis. World J Gastroenterol. 2014 May 7;20(17):4987-93. doi: 10.3748/wjg.v20.i17.4987. PMID 24803810
- [Background] Younossi ZM, Golabi P, de Avila L, Paik JM, Srishord M, Fukui N, Qiu Y, Burns L, Afendy A, Nader F. The global epidemiology of NAFLD and NASH in patients with type 2 diabetes: A systematic review and meta-analysis. J Hepatol. 2019 Oct;71(4):793-801. doi: 10.1016/j.jhep.2019.06.021. Epub 2019 Jul 4. PMID 31279902
- [Background] Harrison SA, Gawrieh S, Roberts K, Lisanti CJ, Schwope RB, Cebe KM, Paradis V, Bedossa P, Aldridge Whitehead JM, Labourdette A, Miette V, Neubauer S, Fournier C, Paredes AH, Alkhouri N. Prospective evaluation of the prevalence of non-alcoholic fatty liver disease and steatohepatitis in a large middle-aged US cohort. J Hepatol. 2021 Aug;75(2):284-291. doi: 10.1016/j.jhep.2021.02.034. Epub 2021 Mar 18. PMID 33746083
- [Background] Allen AM, Therneau TM, Larson JJ, Coward A, Somers VK, Kamath PS. Nonalcoholic fatty liver disease incidence and impact on metabolic burden and death: A 20 year-community study. Hepatology. 2018 May;67(5):1726-1736. doi: 10.1002/hep.29546. Epub 2018 Mar 23. PMID 28941364
- [Background] Chalasani N, Younossi Z, Lavine JE, Charlton M, Cusi K, Rinella M, Harrison SA, Brunt EM, Sanyal AJ. The diagnosis and management of nonalcoholic fatty liver disease: Practice guidance from the American Association for the Study of Liver Diseases. Hepatology. 2018 Jan;67(1):328-357. doi: 10.1002/hep.29367. Epub 2017 Sep 29. No abstract available. PMID 28714183
- [Background] Eslam M, Sanyal AJ, George J; International Consensus Panel. MAFLD: A Consensus-Driven Proposed Nomenclature for Metabolic Associated Fatty Liver Disease. Gastroenterology. 2020 May;158(7):1999-2014.e1. doi: 10.1053/j.gastro.2019.11.312. Epub 2020 Feb 8. PMID 32044314